CLINICAL TRIAL: NCT01668316
Title: Get Active and Eat Right: Moms at Work
Acronym: GEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Greensboro (Other)
Responsible Party: Principal Investigator, Cheryl A Lovelady, PhD RD, Professor, University of North Carolina, Greensboro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM-12-0059
Record Dates: First submitted 2012-08-03; First posted 2012-08-20 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obese; Postpartum; Weight loss; Inflammation; Obesity; Cardiovascular
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Inflammation

ARMS (2):
- Weight loss (Experimental): 12 week weight loss program with biweekly meetings with a Registered Dietitian. Participants will be given a nutrition prescription and asked to record dietary intake online. Participants will be given a pedometer and record daily physical activity.
  Interventions: Behavioral: Weight loss
- Control (No Intervention): Participants asked to not change dietary and physical activity habits.

INTERVENTIONS:
Behavioral: Weight loss — 1. Participants will be prescribed a reduced calorie diet and asked to track their diet three days per week using the online USDA MyPlate SuperTracker. This record will be accessed by the RD in order to provide diet recommendations sent by email.
  2. Participants will be given an exercise prescription, and encouraged to walk briskly with a provided pedometer or exercise at the campus Recreation Center every day. Participants will be asked to record the number of steps and other physical activity in a log book.
  3. Participants will meet with the research staff every other week to measure weight, waist and hip circumference, and record the steps from the pedometer.
  4. Participants will be encouraged to breastfeed their baby and provided with resources for pumping breast milk at work.
  Arms: Weight loss

SUMMARY:
The purpose of this study is to determine the effectiveness of a worksite diet and exercise program on weight loss in postpartum women.

DETAILED DESCRIPTION:
This project is a research study investigating the effects of a worksite diet and exercise intervention on weight loss in overweight postpartum women. Weight loss programs have been shown to be effective in reducing postpartum weight retention. However, high attrition rates in these studies suggest that the added responsibility of a new infant at home and returning to work may limit a woman's ability to follow a diet plan and exercise regularly. We hope that by offering a weight loss program at the workplace, we can increase participant retention and maximize weight loss in this population. Our primary aim is to promote weight loss while preserving lean body mass during the 12 week intervention. Secondary aims include increasing cardiovascular fitness from baseline and improving cardiovascular biomarkers, including total, LDL, and HDL cholesterol, triglycerides, glucose, insulin, and markers of inflammation and metabolism.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older, 10 to 14 weeks postpartum, University faculty, staff, and students, BMI 25-35 or at least 4.5 kilograms heavier than prepregnancy weight, English speaking

Exclusion Criteria:

* Smoking, chronic disease, BMI >35

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-12-21 (Actual); Study Completion 2015-12-21 (Actual)

PRIMARY OUTCOMES:
Weight loss and change in body composition | 12 weeks
  We will be measuring change in weight, waist and hip circumference, and body fat percentage to assess the degree of weight loss and change in body composition at baseline and after the 12 week intervention.

SECONDARY OUTCOMES:
Cholesterol | 12 weeks
  We will be measuring changes in total cholesterol, LDL, and HDL at baseline and after the 12 week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Lovelady, PhD, Principal Investigator — University of North Carolina, Greensboro
Locations (1):
- University of North Carolina at Greensboro, Greensboro, North Carolina, United States